CLINICAL TRIAL: NCT00422604
Title: A Multicentre, Randomised, Partially Blinded, Placebo-controlled, Three-way Crossover, Incomplete Block Design Study to Investigate the Safety, Tolerability, Pharmacodynamics/ Efficacy and Pharmacokinetics of Dual Bronchodilator Therapy With Salmeterol 50µg Twice-daily Plus Two Different Doses of GSK233705B (20 and 50µg Twice-daily), Compared With Placebo, Salmeterol 50µg Twice-daily Alone, and Tiotropium 18µg Once-daily Alone, in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety And Efficacy Of GSK233705 Plus Salmeterol Compared With 2 Active Comparators And Placebo In Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AC2106956
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; plethysmography.; muscarinic receptor antagonist; anticholinergic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: salmeterol
Drug: tiotropium
Drug: GSK233705
  Other Names: salmeterol; tiotropium

SUMMARY:
The safety, tolerability, pharmacokinetics and pharmacodynamics/efficacy profiles of two different doses of GSK233705 will be compared with 2 active comparators and placebo, all medication delivered via dry powder inhaler.

DETAILED DESCRIPTION:
A multi-centre, randomised, partially blinded, placebo-controlled, three-way crossover, incomplete block design study to investigate the, safety, tolerability, pharmacodynamics/efficacy and pharmacokinetics of dual bronchodilator therapy with salmeterol 50 mcg twice daily plus two different doses of GSK233705 (20 and 50 mcg twice daily), compared with placebo, salmeterol 50 mcg twice daily alone, and tiotropium 18 mcg once daily alone, in subjects with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion criteria:

* females of non-childbearing potential or postmenopausal;
* history of COPD as defined by ATS/ERS criteria;
* moderate COPD responsive to ipratropium and salbutamol;
* current smoker or ex-smoker.

Exclusion criteria:

* no instable COPD; max 1000 mcg inhaled steroids per day; no B-blockers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Bronchodilator effect of GSK233705 plus salmeterol at day 7, compared with placebo in COPD subjects.

SECONDARY OUTCOMES:
Bronchodilator effect of salmeterol alone and tiotropium alone compared with placebo and GSK233705 at day 7. Safety and tolerability of GSK233705 plus salmeterol and the 2 active comparators at day 7.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- GSK Investigational Site, Helsinki, Finland
- Germany (2):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- Netherlands (4):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Veldhoven
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- United Kingdom (2):
  - GSK Investigational Site, Upton Road, Slough, Berkshire
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Beier J, van Noord J, Deans A, Brooks J, Maden C, Baggen S, Mehta R, Cahn A. Safety and efficacy of dual therapy with GSK233705 and salmeterol versus monotherapy with salmeterol, tiotropium, or placebo in a crossover pilot study in partially reversible COPD patients. Int J Chron Obstruct Pulmon Dis. 2012;7:153-64. doi: 10.2147/COPD.S26100. Epub 2012 Mar 5. PMID 22419863
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2106956 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register